CLINICAL TRIAL: NCT00177957
Title: Gram Negative Bacteremia, Risk Factors for Failure of Therapy
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: PI discretionary funding (Unknown)
Responsible Party: Principal Investigator, Yohei Doi, Associate Professor, University of Pittsburgh
Other Study IDs: IRB # 0504090
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Gram-Negative Bacterial Infections
Keywords: Gram negative bacteremia
MeSH Terms: conditions — Gram-Negative Bacterial Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aims of this study are to:

* Determine the risk factors for multidrug resistance in bloodstream isolates of Gram negative bacilli
* Determine the mechanisms of multidrug resistance in bloodstream isolates of Gram negative bacilli
* Determine the risk factors for failure of prompt clearance of the blood of Gram negative bacteria
* Determine the survival of patients with Gram negative bacteremia
* Determine if failure of prompt clearance of the blood of Gram negative bacteria is a predictor of mortality following this infection

DETAILED DESCRIPTION:
The following variables will be followed: time and location of positive cultures, underlying diseases and severity of illness, recent immunomodulative therapies, physical exam findings, laboratory and radiographical data, antimicrobial usage within 14 days of onset of bacteremia, microbiological data and resistance patterns, choice of antibiotics once organism identified, suspected source of bacteremia, bacteriological outcomes, laboratory results, demographic information, medications, clinical outcome,gender, height, weight, ethnicity, and past medical history (please see attached clinical data collection worksheet dated 4/2005). We will also collect information retrospectively for one year and prospectively for one year. The bacteria in the patient's blood cultures will be subcultured (after the diagnosis has been obtained since the microbiology lab would otherwise destroy the culture) and provided to the honest broker who will deidentify the specimen and link it to the medical information collected (which will also be deidentified by the honest broker). The following evaluation will be performed on these samples. The minimal inhibitory concentration of the antibiotic used in treatment will be performed by the E-Test method (AB Biodisk, Solna, Sweden). Specific mechanisms of antimicrobial resistance will be studied with emphasis on the presence of beta-lactamases produced by the bacteria. This evaluation will be performed by analytical isoelectric focusing techniques as well as PCR and gene sequencing analysis to determine genes encoding beta-lactamases. Biologic samples will be under the control of the principal investigator of this research project. All samples provided to the investigators are deidentified by the honest broker and will be coded with numbers. The information linking these code numbers to the corresponding subjects' identities will be kept in a separate, secure location that only the honest broker has access to. The investigators on this study will keep the samples indefinitely. Samples will be kept in the investigator's laboratory located in Scaife Hall, room 812, 3500 Terrace Street. At no time with the research investigators have access to any patient identifiers.

ELIGIBILITY:
Inclusion Criteria:

* All patients at the aforementioned institutions that have Gram negative bacteremia will be included in the study.
* Women with childbearing potential will also be included in this study. Since this is an observational study, no added risk is conferred to the woman or potential progeny. HIV serostatus will not be specifically investigated for participation in this study.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with gram negative bacteremia
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2005-04; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
outcome of dead or alive post treatment | December 2020
  dead or alive

CONTACTS AND LOCATIONS:
Overall Officials: Yohei Doi, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
not sharing